CLINICAL TRIAL: NCT06634589
Title: A Phase 1b/2, Open-Label, Master Protocol Study of BTK-Degrader BGB-16673 in Combination With Other Agents in Patients With Relapsed or Refractory B-Cell Malignancies
Brief Title: A Study to Investigate Safety and Effectiveness of BGB-16673 in Combination With Other Agents in Participants With Relapsed or Refractory B-Cell Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BeOne Medicines (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-16673-104; 2024-516234-35-00 (EU CTIS Number); CTR20244676 (Registry Identifier: ChinaDrugTrials)
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: B-cell Malignancy; Relapsed Cancer; Refractory Cancer; B-cell Lymphoma
Keywords: R/R B-Cell Malignancies; relapsed or refractory B-Cell Malignancies; B-Cell malignancy; BGB-16673; sonrotoclax; zanubrutinib; B-cell lymphoma; Bruton Tyrosine Kinase (BTK); Mosunetuzumab; Glofitamab
MeSH Terms: conditions — Recurrence; Neoplasms; Lymphoma, B-Cell | interventions — zanubrutinib; glofitamab; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Substudy 1 Part 1a: Dose Escalation (Experimental): Sequential cohorts of increasing dose level combinations of BGB-16673 and sonrotoclax will be evaluated in participants with selected B-cell malignancies.
  Interventions: Drug: BGB-16673; Drug: Sonrotoclax
- Substudy 1 Part 1b: Safety Expansion (Experimental): Cohorts of select dose level combinations of BGB-16673 and sonrotoclax will be evaluated in participants with selected B-cell malignancies.
  Interventions: Drug: BGB-16673; Drug: Sonrotoclax
- Substudy 2 Part 1a: Dose Escalation (Experimental): Sequential cohorts of increasing dose level combinations of BGB-16673 and zanubrutinib will be evaluated in participants with selected B-cell malignancies.
  Interventions: Drug: BGB-16673; Drug: Zanubrutinib
- Substudy 2 Part 1b: Safety Expansion (Experimental): Cohorts of select dose level combinations of BGB-16673 and zanubrutinib will be evaluated in participants with selected B-cell malignancies.
  Interventions: Drug: BGB-16673; Drug: Zanubrutinib
- Substudy 3 Part 1a: Dose Escalation (Experimental): Sequential cohorts of increasing dose level combinations of BGB-16673 and mosunetuzumab will be evaluated in participants with selected B-cell malignancies.
  Interventions: Drug: BGB-16673; Drug: Mosunetuzumab
- Substudy 3 Part 1b: Safety Expansion (Experimental): Cohorts of select dose level combinations of BGB-16673 and mosunetuzumab will be evaluated in participants with selected B-cell malignancies.
  Interventions: Drug: BGB-16673; Drug: Mosunetuzumab
- Substudy 4 Part 1a: Dose Escalation (Experimental): Sequential cohorts of increasing dose level combinations of BGB-16673 and glofitamab will be evaluated in participants with selected B-cell malignancies. Participants will receive obinutuzumab as pretreatment prior to the start of combination treatment.
  Interventions: Drug: BGB-16673; Drug: Glofitamab; Drug: Obinutuzumab
- Substudy 4 Part 1b: Safety Expansion (Experimental): Cohorts of select dose level combinations of BGB-16673 and glofitamab will be evaluated in participants with selected B-cell malignancies.
  Interventions: Drug: BGB-16673; Drug: Glofitamab; Drug: Obinutuzumab

INTERVENTIONS:
Drug: BGB-16673 — Administered orally
Drug: Sonrotoclax — Administered orally
  Other Names: BGB-11417
  Arms: Substudy 1 Part 1a: Dose Escalation; Substudy 1 Part 1b: Safety Expansion
Drug: Zanubrutinib — Administered orally
  Arms: Substudy 2 Part 1a: Dose Escalation; Substudy 2 Part 1b: Safety Expansion
Drug: Mosunetuzumab — Administered subcutaneously
  Arms: Substudy 3 Part 1a: Dose Escalation; Substudy 3 Part 1b: Safety Expansion
Drug: Glofitamab — Administered intravenously
  Arms: Substudy 4 Part 1a: Dose Escalation; Substudy 4 Part 1b: Safety Expansion
Drug: Obinutuzumab — Administered intravenously
  Arms: Substudy 4 Part 1a: Dose Escalation; Substudy 4 Part 1b: Safety Expansion

SUMMARY:
The purpose of this study is to measure the safety, preliminary antitumor activity, pharmacokinetics, and pharmacodynamics with BGB-16673 in combination with other agents in participants with relapsed or refractory (R/R) B-cell malignancies. This study is structured as a master protocol with separate substudies. This study currently includes four substudies, and more substudies may be added as other combination agents are identified.

DETAILED DESCRIPTION:
This new study will check how safe and helpful a potential anticancer drug called BGB-16673 is in participants with R/R B-cell malignancies when it is given in combination with other medicines - sonrotoclax in substudy 1, zanubrutinib in substudy 2, mosunetuzumab in substudy 3, and glofitamab in substudy 4.

Our company, previously known as BeiGene, is now officially BeOne Medicines. Because some of our older studies were sponsored under the name BeiGene, you may see both names used for this study on this website.

ELIGIBILITY:
Key Inclusion Criteria:

* Must sign the informed consent form (ICF) and be capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the ICF
* Confirmed diagnosis of a R/R B-cell malignancy
* Protocol-defined measurable disease
* Stable Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2
* Adequate organ function
* Female participants of childbearing potential must be willing to use a highly effective method of birth control and refrain from egg donation for the duration of the study and for 30 days after the last dose of BGB-16673 or zanubrutinib, 60 days after the last dose of glofitamab, or 90 days after the last dose of sonrotoclax or mosunetuzumab. A negative urine or serum pregnancy test result must be provided 10-14 days before the first dose of study treatment
* Nonsterile male participants must be willing to use a highly effective method of birth control and refrain from sperm donation for the duration of the study and for 30 days after the last dose of BGB-16673 or zanubrutinib, 60 days after the last dose of glofitamab, or 90 days after the last dose of sonrotoclax or mosunetuzumab
* Substudies 1, 3, and 4 Inclusion Criterion:

  * Adequate renal function as indicated by estimated glomerular filtration rate (eGFR) of ≥ 50 mL/min
* Substudy 2 Inclusion Criteria:

  * Bruton tyrosine kinase (BTK) inhibitor-naive, or previously received treatment with a covalent BTK inhibitor and discontinued for reasons other than clinical progression
  * Adequate renal function as indicated by eGFR of ≥ 30 mL/min

Key Exclusion Criteria:

* Treatment-naive B-cell malignancies
* Unable to comply with the requirements of the protocol
* Active leptomeningeal disease or uncontrolled, untreated brain metastasis
* Any malignancy ≤ 2 years before first dose of study treatment except for the specific cancer under investigation in this study or any locally recurring cancer that has been treated curatively
* Autologous stem cell transplant ≤ 3 months prior to screening or chimeric antigen T-cell therapy ≤ 3 months prior to screening
* Substudies 1 and 2: Prior allogeneic stem cell transplant with active graft-versus-host disease (GVHD), or requiring immunosuppressive drugs for treatment of GVHD, or who have taken calcineurin inhibitors within 4 weeks prior to consent
* Participants who have a history of severe allergic reactions or hypersensitivity to the active ingredient and excipients of BGB-16673, sonrotoclax, zanubrutinib, mosunetuzumab, or glofitamab
* Substudy 1 Exclusion Criterion:

  * Prior treatment with a B-cell lymphoma-2 (Bcl-2) inhibitor (with exception for participants who relapsed ≥ 24 months after completion of a full course of a prior Bcl-2 inhibitor containing regimen)
* Substudy 2 Exclusion Criterion:

  * Participants who discontinued prior zanubrutinib treatment due to intolerance
* Substudies 3 and 4 Exclusion Criteria:

  * Prior exposure to a CD20 x CD3 T-cell engager antibody treatment
  * All participants with a prior allogeneic stem cell transplant

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2028-12-02 (Estimated); Study Completion 2029-12-02 (Estimated)

PRIMARY OUTCOMES:
Substudy 1 Part 1a: Number of participants with dose-limiting toxicities (DLTs), treatment-emergent adverse events, treatment-related adverse events, and serious adverse events | From the first dose of study drug(s) to 30 days after the last dose; up to approximately 2 years
Substudy 1 Part 1b: Number of participants with treatment-emergent adverse events, treatment-related adverse events, and serious adverse events | From the first dose of study drug(s) to 30 days after the last dose; up to approximately 2 years
Substudy 2 Part 1a: Number of participants with dose-limiting toxicities (DLTs), treatment-emergent adverse events, treatment-related adverse events, and serious adverse events | From the first dose of study drug(s) to 30 days after the last dose; up to approximately 2 years
Substudy 2 Part 1b: Number of participants with treatment-emergent adverse events, treatment-related adverse events, and serious adverse events | From the first dose of study drug(s) to 30 days after the last dose; up to approximately 2 years
Substudy 3 Part 1a: Number of participants with dose-limiting toxicities (DLTs), treatment-emergent adverse events, treatment-related adverse events, and serious adverse events | From the first dose of study drug(s) to 30 days after the last dose; up to approximately 2 years
Substudy 3 Part 1b: Number of participants with treatment-emergent adverse events, treatment-related adverse events, and serious adverse events | From the first dose of study drug(s) to 30 days after the last dose; up to approximately 2 years]
Substudy 4 Part 1a: Number of participants with dose-limiting toxicities (DLTs), treatment-emergent adverse events, treatment-related adverse events, and serious adverse events | From the first dose of study drug(s) to 30 days after the last dose; up to approximately 2 years
Substudy 4 Part 1b: Number of participants with treatment-emergent adverse events, treatment-related adverse events, and serious adverse events | From the first dose of study drug(s) to 30 days after the last dose; up to approximately 2 years

SECONDARY OUTCOMES:
Substudy 1 Parts 1a and 1b: Overall Response Rate (ORR) in participants with B-cell malignancies | Up to approximately 3 years
  ORR is defined as the percentage of participants with complete response (CR) or partial response (PR) as assessed by investigator.
Substudy 1 Parts 1a and 1b: Duration of Response (DOR) | Up to approximately 3 years
  DOR is defined as the time from the first documented response to documented disease progression or death, whichever occurs first.
Substudy 1 Parts 1a and 1b: Time to Response (TTR) | Up to approximately 3 years
  TTR is defined as the time from treatment initiation to first documented response.
Substudy 1 Part 1a: Area under the plasma concentration-time curve (AUC) of BGB-16673 and sonrotoclax | From Week 1 to Week 17
Substudy 1 Part 1a: Maximum observed concentration (Cmax) of BGB-16673 and sonrotoclax | From Week 1 to Week 17
Substudy 1 Part 1a: Time to maximum concentration (Tmax) of BGB-16673 and sonrotoclax | From Week 1 to Week 17
Substudy 1 Part 1a: Terminal half-life (t1/2) of BGB-16673 and sonrotoclax | From Week 1 to Week 17
Substudy 1 Parts 1a and 1b: Trough concentration (Ctrough) of BGB-16673 and sonrotoclax | From Week 1 to Week 17
Substudy 1 Part 1b: Number of patients with complete response or complete response with incomplete count recovery (CR/CRi) who achieve undetectable minimal residual disease (uMRD) | Up to approximately 3 years
Substudy 2 Parts 1a and 1b: ORR in participants with B-cell malignancies | Up to approximately 3 years
  ORR is defined as the percentage of participants with complete response (CR) or partial response (PR) as assessed by the investigator.
Substudy 2 Parts 1a and 1b: DOR | Up to approximately 3 years
  DOR is defined as the time from the first documented response to documented disease progression or death, whichever occurs first.
Substudy 2 Parts 1a and 1b: TTR | Up to approximately 3 years
  TTR is defined as the time from treatment initiation to the first documented response.
Substudy 2 Part 1a: Area under the plasma concentration-time curve (AUC) of BGB-16673 and zanubrutinib | From Week 1 to Week 17
Substudy 2 Part 1a: Maximum observed concentration (Cmax) of BGB-16673 and zanubrutinib | From Week 1 to Week 17
Substudy 2 Part 1a: Time to maximum concentration (Tmax) of BGB-16673 and zanubrutinib | From Week 1 to Week 17
Substudy 2 Part 1a: Terminal half-life (t1/2) of BGB-16673 and zanubrutinib | From Week 1 to Week 17
Substudy 2 Parts 1a and 1b: Trough concentration (Ctrough) of BGB-16673 and zanubrutinib | From Week 1 to Week 17 for Part 1a; From Week 1 to Week 5 for Part 1b
Substudy 3 Parts 1a and 1b: ORR in participants with B-cell malignancies | Up to approximately 3 years
  ORR is defined as the percentage of participants with complete response (CR) or partial response (PR) as assessed by the investigator.
Substudy 3 Parts 1a and 1b: DOR | Up to approximately 3 years
  DOR is defined as the time from the first documented response to documented disease progression or death, whichever occurs first.
Substudy 3 Parts 1a and 1b: TTR | Up to approximately 3 years
  TTR is defined as the time from treatment initiation to the first documented response.
Substudy 3 Part 1a: Area under the plasma concentration-time curve (AUC) of BGB-16673 and mosunetuzumab | From Week 1 to Week 12
Substudy 3 Part 1a: Maximum observed concentration (Cmax) of BGB-16673 and mosunetuzumab | From Week 1 to Week 12
Substudy 3 Part 1a: Time to maximum concentration (Tmax) of BGB-16673 and mosunetuzumab | From Week 1 to Week 12
Substudy 3 Part 1a: Terminal half-life (t1/2) of BGB-16673 and mosunetuzumab | From Week 1 to Week 12
Substudy 3 Parts 1a and 1b: Trough concentration (Ctrough) of BGB-16673 and mosunetuzumab | From Week 1 to Week 36
Substudy 4 Parts 1a and 1b: ORR in participants with B-cell malignancies | Up to approximately 3 years
  ORR is defined as the percentage of participants with partial response (PR) or better as assessed by the investigator.
Substudy 4 Parts 1a and 1b: DOR | Up to approximately 3 years
  DOR is defined as the time from the first documented response to documented disease progression or death, whichever occurs first.
Substudy 4 Parts 1a and 1b: TTR | Up to approximately 3 years
  TTR is defined as the time from treatment initiation to the first documented response.
Substudy 4 Part 1a: Area under the plasma concentration-time curve (AUC) of BGB-16673 | From Week 1 to Week 10
Substudy 4 Part 1a: Maximum observed concentration (Cmax) of BGB-16673 | From Week 1 to Week 10
Substudy 4 Part 1a: Time to maximum concentration (Tmax) of BGB-16673 | From Week 1 to Week 10
Substudy 4 Part 1a: Terminal half-life (t1/2) of BGB-16673 | From Week 1 to Week 10
Substudy 4 Parts 1a and 1b: Trough concentration (Ctrough) of BGB-16673 | From Week 1 to Week 10

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeOne Medicines
Locations (41):
- United States (17):
  - Mayo Clinic Phoenix, Phoenix, Arizona
  - University of Southern Californianorris Comprehensive, Los Angeles, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - The University of Kansas Cancer Center, Westwood, Kansas
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Summit Medical Group, Florham Park, New Jersey
  - Icahn School of Medicine At Mount Sinai, New York, New York
  - Weill Cornell Medical College Newyork Presbyterian Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center Mskcc, New York, New York
  - University of Rochester, Rochester, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - The University of Texas Md Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Wisconsin, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (6):
  - St George Hospital, Kogarah, New South Wales
  - Mater Cancer Care Centre, South Brisbane, Queensland
  - Monash Health, Clayton, Victoria
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
- China (5):
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Sun Yat Sen University Cancer Center, Guangzhou, Guangdong
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital, Zhejiang University School of Medicinechengzhan, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
- Germany (3):
  - Universitatsklinikum Carl Gustav Carus An Der Technischen Universitat Dresden, Dresden
  - Universitatsklinikum Jena Klinik Fur Innere Medizin Ii, Jena
  - Universitaetsklinikum Ulm, Ulm
- Italy (4):
  - Azienda Ospedaliera Universitaria Policlinico Santorsola Malpighi, Bologna
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
  - Istituto Nazionale Tumori Fondazione G Pascale, Napoli
  - Centroricerche Cliniche Di Verona Srl, Verona
- New Zealand (2):
  - North Shore Hospital, Auckland
  - Auckland City Hospital, Auckland
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Szpital Kliniczny Mswia Z Warmisko Mazurskim Centrum Onkologii, Olsztyn
  - Szpital Wojewodzki W Opolu Sp Z Oo Oddzia Hematologii I Onkologii Hematologicznej, Opole
  - Narodowy Instytut Onkologii Im Marii Sklodowskiej Curie Hematology Unit, Warsaw

IPD SHARING:
Plan to Share IPD: Yes
BeOne shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeOne shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeOne review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beonemedicines.com/science/clinical-trials/